CLINICAL TRIAL: NCT01425749
Title: T Cell Activation and Immune Cell Function in Melanoma Patients Treated With recMAGE-A3 + AS15 Immunological Adjuvant System
Brief Title: Study to Assess Safety and Immune Response of Stage IIB-IV Resected Melanoma After Treatment With MAGE-A3 ASCI
Acronym: Mel55
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery; Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSlingluff
Record Dates: First submitted 2011-07-19; First posted 2011-08-30 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Melanoma
Keywords: melanoma; MAGE-A3; immunotherapy; adjuvant; skin cancer; skin diseases; immunology
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Intramuscular injections of recMAGE-A3 + AS15 ASCI.
  Interventions: Biological: recMAGE-A3 + AS15 ASCI
- Arm B (Experimental): Intradermal/Subcutaneous injections of recMAGE-A3 + AS15 ASCI. Requires an injection site biopsy at Day 8 and Day 50.
  Interventions: Biological: recMAGE-A3 + AS15 ASCI

INTERVENTIONS:
Biological: recMAGE-A3 + AS15 ASCI — Injections of recMAGE-A3 + AS15 ASCI will be given 5 times at 3-week intervals. This will either be administered cutaneously or intramuscularly depending on the study group. The injected doses will be administered in alternating extremities at each visit.
  Other Names: recMAGE-A3 + AS15 ASCI IM; recMAGE-A3 + AS15 ASCI ID/SC

SUMMARY:
The goals of this study are to 1) assess the safety of recombinant MAGE-A3 protein combined with AS15 Immunological Adjuvant System (recMAGE-A3 + AS15) as an Antigen-Specific Cancer Immunotherapeutic (MAGE-A3 ASCI) when administered in two different administration sites, intramuscular (IM) or intradermal/subcutaneous (ID/SC), and 2) to provide preliminary data on the immunological response to ASCI in the injection site microenvironment, in the node draining the vaccine site (sentinel immunized node) and in the blood and whether there are large differences in the magnitude, persistence, or type of immune response induced as a function of the ASCI injection. Evaluation of immune responses to the ASCI will include, amonth others antiMAGE-A3 antibody responses and CD4+ and CD8+ T cell responses.

DETAILED DESCRIPTION:
This was an open-label randomized single institution pilot study to evaluate the safety and immunologic response to MAGE-A3 immunotherapeutic administered by either of two injection routes (i.m. or i.d./s.c.). Patients were studied following IRB approval (IRB #15398) and documentation of informed consent. The trial was registered in clinicaltrials.gov (NCT01425749), and was performed at the University of Virginia.

MAGE-A3 immunotherapeutic (0.5 ml) was administered five times (weeks 0, 3, 6, 9, 12) in extremities uninvolved with melanoma. Vaccines 1 and 3 were administered at the same site: other vaccine sites were rotated among available extremities. Subjects were randomized 1:1, within each stratum (AJCC stage II/III or IV), to i.m. (Group A) or i.d./s.c. (Group B) administration. The randomization code was generated by the study statistician using varying block sizes of 2 to 4. For group B patients, half of the dose was injected s.c., then the needle was withdrawn to the dermis, then advanced intradermally from that same puncture site and the remaining half dose was injected i.d. Immune responses were evaluated in a SIN and PBMC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven melanoma that meets one of the following two criteria:

  * Stage IIB-IV melanoma rendered clinically free of disease by surgery, other therapy, or spontaneous remission within 6 months prior to registration.
  * Stage III or IV melanoma with disease. Patients may be eligible if there are definite or equivocal findings of persistent or metastatic disease as long as those findings do not meet RECIST criteria for measurable disease.
* Expression of MAGE-A3 by the tumor (primary or metastasis).
* Patients may have had multiple primary melanomas.
* Patients may have had, or may have, a metastasis from a cutaneous, mucosal, unknown primary site.
* Patients with brain metastases may be eligible if all of the following are true:

  * The total number of brain metastases ever is less than or equal to 3.
  * The brain metastases have been completely removed by surgery or have been treated completely by stereotactic radiotherapy. Stereotactic radiotherapy, such as gamma knife, can be used up to 1 week prior to study entry.
  * There has been no evident growth of any brain metastasis since treatment.
  * No treated brain metastasis is greater than 2 cm in diameter at the time of protocol entry.
* Patients must have at least two intact axillary and/or inguinal lymph node basins.
* The interferon education packet must be completed satisfactorily for those who are eligible for, but refuse, interferon therapy.
* All patients must have:

  * ECOG performance status of 0 or 1.
  * Ability and willingness to give informed consent.
* Laboratory parameters as follows:

  1. ANC > 1000/mm3, and Platelets > 75,000/mm3 and Hgb > 9 g/dL
  2. Hepatic:

     AST and ALT up to 2.5 x upper limits of normal (ULN) Bilirubin up to 2.5 x ULN Alkaline phosphatase up to 2.5 x ULN LDH up to 2x ULN
  3. Renal:

     Creatinine up to 1.5 x ULN
  4. Serology:

     HIV negative (antibody screening), Hepatitis C negative
  5. HGBA1C level of < 7.5%
* Patients must be 18 years or older at study entry

Exclusion Criteria:

* Patients with primary ocular melanoma.
* Patients who have had brain metastases unless they meet the criteria outlined in the inclusion criteria
* Patients who are currently receiving systemic cytotoxic chemotherapy, radiation, monoclonal antibody therapy, or other experimental therapy, or who have received this therapy within the preceding 4 weeks. Patients who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks.
* Patients who have received isolated limb infusion (ILI) or isolated limb perfusion (ILP) for melanoma will not be eligible unless they have experienced tumor progression after the ILI/ILP, and the ILI/ILP was not performed within the prior 12 weeks.
* Patients will not be eligible if there is clinically detectable melanoma deemed likely by the investigator to require intervention during the first 12 weeks of the study that would require premature discontinuation.
* Patients with known or suspected allergies to any component of the MAGE-A3 ASCI.
* Patients receiving the following medications at study entry or within the preceding 4 weeks are excluded, except as specified below:

  1. Agents with putative immunomodulating activity, but with the exception of non-steroidal anti-inflammatory agents and topical steroids.
  2. Antibodies to CTLA-4, PD-1, PD-L1, or CD137 may not have been received in the past 12 weeks, and patients will be eligible only if there has been melanoma progression since that therapy was administered.
  3. Allergy desensitization injections.
  4. Systemic corticosteroids, administered parenterally or orally. Inhaled steroids are not permitted. Topical corticosteroids are acceptable, including steroids with very low solubility administered nasally for local effects only.
  5. Any growth factors (e.g. GM-CSF, G-CSF, erythropoietin).
  6. Interferon therapy.
  7. Interleukin-2 or other interleukins.
  8. Targeted therapies designed to inhibit BRAF, MAPKinase, mTOR, or their signaling pathways.
* Prior active immunotherapy or vaccines for melanoma may be an exclusion criterion in some circumstances. Exceptions to this exclusion criterion are as follows:

  1. Patients who have recurred or progressed either after or during administration of a melanoma vaccine may be eligible to enroll in this study 12 weeks following their last vaccination.
  2. Patients may not have been previously administered the synthetic MAGE-A3 protein, though prior vaccinations with up to 4 synthetic MAGE-A3 peptides (up to 16 amino acids in length, each) is allowed.
* Pregnancy or the possibility of becoming pregnant during vaccine administration. Female patients of child-bearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the first MAGE-A3 ASCI dose. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. Women must also not be breast feeding. This is consistent with existing standards of practice for vaccine and chemotherapy protocols.
* Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
* Patients classified according to the New York Heart Association classification as having Class III or IV heart disease.
* Patients with a body weight < 110 lbs because of the amount and frequency with which blood will be drawn, and because of the biopsies required.
* Patients must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Patients with an active autoimmune disorder requiring these therapies are also excluded. The following will not be exclusionary:

  * Laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring NSAID medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Slingluff CL Jr, Petroni GR, Olson WC, Smolkin ME, Chianese-Bullock KA, Mauldin IS, Smith KT, Deacon DH, Varhegyi NE, Donnelly SB, Reed CM, Scott K, Galeassi NV, Grosh WW. A randomized pilot trial testing the safety and immunologic effects of a MAGE-A3 protein plus AS15 immunostimulant administered into muscle or into dermal/subcutaneous sites. Cancer Immunol Immunother. 2016 Jan;65(1):25-36. doi: 10.1007/s00262-015-1770-9. Epub 2015 Nov 18. PMID 26581199

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Intramuscular Injections: Intramuscular injections.
  recMAGE-A3 + AS15 ASCI: Injections will be given 5 times at 3-week intervals. This will either be administered cutaneously or intramuscularly depending on the study group. The injected doses will be administered in alternating extremities at each visit.
- Arm B: Intradermal/Subcutaneous Injections: Intradermal/Subcutaneous injections. Requires an injection site biopsy at Day 8 and Day 50.
  recMAGE-A3 + AS15 ASCI: Injections will be given 5 times at 3-week intervals. This will either be administered cutaneously or intramuscularly depending on the study group. The injected doses will be administered in alternating extremities at each visit.
Period: Overall Study
Arm/Group | Arm A: Intramuscular Injections | Arm B: Intradermal/Subcutaneous Injections
Started | 13 | 12
Completed | 13 | 11
Not Completed | 0 | 1
Not completed — progression of melanoma | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Intramuscular injections.
  recMAGE-A3 + AS15 ASCI: Injections will be given 5 times at 3-week intervals. This will either be administered cutaneously or intramuscularly depending on the study group. The injected doses will be administered in alternating extremities at each visit.
- Arm B: Intradermal/Subcutaneous injections. Requires an injection site biopsy at Day 8 and Day 50.
  recMAGE-A3 + AS15 ASCI: Injections will be given 5 times at 3-week intervals. This will either be administered cutaneously or intramuscularly depending on the study group. The injected doses will be administered in alternating extremities at each visit.
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Full Range); unit: years] | 56 [39 to 82] | 54 [40 to 69] | 55 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Stage of Melanoma [Number; unit: participants] — AJCC staging, version 7
  participants
    Stage IIIB | 3 | 5 | 8
    Stage IIIC | 5 | 3 | 8
    Stage IV | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as a Measure of Safety and Tolerability
Description: grade 2 treatment-related adverse events graded by CTCAE v4
Time Frame: Over 6 months
Population: All eligible patients.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 13 | 12
participants
  Chills | 1 | 0
  Fatigue | 4 | 2
  Fever | 1 | 0
  Flu-like symptoms | 1 | 2
  Injection site reaction | 10 | 7
  Wound complication | 0 | 1
  lymphocyte count decreased | 1 | 0
  grade 3 or higher adverse events | 0 | 0

2. Primary Outcome: Enumeration of CD4 and CD8 T Cell Responses to MAGE-A3 Epitopes in the Injection Site-draining Lymph Node (Sentinel Immunized Node, SIN) as a Measure of Immunogenicity.
Description: Flow cytometry on in vitro stimulated lymphocytes. A positive immune response was identified as one with bifunctional CD4+ or CD8+ T cells, producing both TNF alpha and IFN-gamma after exposure to antigen.
Time Frame: One week after 3 doses of study drug, on day 22.
Population: Eligible participants with evaluable sentinel immunized node specimens.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 13 | 11
participants
  CD4+ T cell response | 4 | 7
  CD8+ T cell response | 0 | 1

3. Secondary Outcome: Enumeration of CD4+ and CD8+ T Cells Reactive to MAGE-A3 Epitopes in Peripheral Blood as a Measure of Immunogenicity.
Description: The analysis determined the proportion of CD4+ (and/or CD8+) T cells producing IFN-gamma or TNFα, or both, in response to MAGE-A3 peptide pools (with irrelevant peptide as negative control). T cell response was defined when T cells producing both IFNγ and TNFα in response to MAGE-A3 peptides exceeded (a) twice the maximum of 2 negative controls (PRAME peptides, media only), corrected for pre-existing response; and (b) exceeded the negative controls by at least 0.2% of the T cell population. These criteria also were used to define immunogenicity by ELIspot (IFNγ only). If the negative control values for a given sample were zero, a meaningful fold-increase could not be calculated; so, in those cases, we used the minimum detectable value among all similar assays (0.06%) as the negative control value for that sample.
Time Frame: Over 6 months
Population: All eligible patients with evaluable peripheral blood mononuclear cells; this corresponds to all enrolled patients.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 13 | 12
participants
  CD4+ T cell response | 4 | 6
  CD8+ T cell response | 1 | 2

4. Secondary Outcome: Identification of Antibody Responses to MAGE-A3 After MAGE-A3 ASCI Administration as a Measure of Immunogenicity.
Description: Antibody responses were assessed in serum by ELISA, assay for IgG. Seroconversion was defined as a detectable Ab response by ELISA (>20 EU/ml).
Time Frame: Over 6 months, typically weeks 1, 7, 13, 26
Population: All eligible participants.
Measure: Number; unit: percentage of evaluable participantes
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 13 | 12
percentage of evaluable participantes
  Seropositivity week 0 | 8 | 0
  Seropositivity week 1 | 38 | 8
  Seropositivity week 7 | 100 | 100
  Seropositivity week 13 | 100 | 100
  Seropositivity week 26 | 100 | 100

5. Secondary Outcome: Characterization of the Maturation and Activation of Dendritic Cell (DC) Populations in the Sentinel Immunized Node (SIN) After Treatment With MAGE-A3 ASCI.
Description: Number of CD83+ cells (mature DC) and CD1a+ cells (immature DC/Langerhans cells) per mm^2 in cross-sections of sentinel immunized nodes
Time Frame: Over 3 weeks
Population: Evaluable patients with sufficient node sample for the analysis of DC infiltrates.
Measure: Mean (Standard Deviation); unit: cells per mm^2 in SIN
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 11 | 11
cells per mm^2 in SIN
  CD83+ cells | 10 (14) | 9 (13)
  CD1a+ | 42 (33) | 28 (21)

6. Secondary Outcome: A Preliminary Evaluation of Cellular Components of the Injection Site Microenvironment for Cutaneous Immunization With MAGE-A3 ASCI (Activated T Cells, Th1,Th2, Th17 Infiltrating CD4 Cells, Regulatory T Cells, and Myeloid-derived Suppressor Cells).
Description: Cells per mm^2 in the superficial dermis at the vaccine site microenvironment, by enumeration of immunohistochemically stained slides. Biopsies of the vaccine sites were taken at week 1 (1 week after the first vaccine) and week 7 (1 week after the 3rd vaccine). This only was evaluable in Arm B patients.
Time Frame: Over 6 months
Population: Participants enrolled on Arm B who had sufficient biopsy site samples.
Measure: Mean (Standard Deviation); unit: cells per mm^2 of dermis
Arm/Group | Arm B
Number analyzed (Participants) | 11
cells per mm^2 of dermis
  CD8 T cells, week 1 | 129 (81.6)
  CD4 T cells, week 1 | 203.6 (168.8)
  CD1a+ cells, week 1 | 10.9 (13.8)
  CD83+ cells, week 1 | 12.6 (13.7)
  FoxP3+ cells, week 1 | 43.6 (63.3)
  Tbet+ cells, week 1 | 53 (80.4)
  GATA3+ cells, week 1 | 85.6 (73.2)
  RORgamma-t + cells, week 1 | 28 (46.3)
  CD20+ cells, week 1 | 3.9 (2.9)
  Eosinophils, week 1 | 0.0 (0.0)
  CD8+ T cells, week 7 | 99.9 (56.9)
  CD4+ T cells, week 7 | 125.9 (103.1)
  CD1a+ cells, week 7 | 9 (8.5)
  CD83+ cells, week 7 | 7.8 (6.7)
  FoxP3+ cells, week 7 | 28.5 (21)
  Tbet+ cells, week 7 | 14.1 (8.5)
  GATA3+ cells, week 7 | 41.3 (21.1)
  RORgammat+ cells, week 7 | 7.8 (6.1)
  CD20+ cells, week 7 | 6.5 (7.1)
  Eosinophils, week 7 | 0.1 (0.2)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Treatment-related adverse events (AEs) were recorded. At each clinic visit, each patient was completely evaluated by a licensed clinician, for physical exam and history and review of toxicity diaries. Additional AEs were captured from laboratory tests. Grade 2 AEs are listed under primary endpoint. AEs of grade 3 or higher are reported here (none).
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=13) | Arm B (N=12)
Diarrhea (Gastrointestinal disorders) | 2 | 1
Mucositis Oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 3
Chills (General disorders) | 9 | 4
Fatigue (General disorders) | 12 | 12
Fever (General disorders) | 4 | 5
Flu-like symptoms (General disorders) | 6 | 7
injection site reaction (General disorders) | 13 | 12
localized edema (General disorders) | 0 | 1
other (General disorders) | 1 | 0
Autoimmune disorder (General disorders) | 2 | 1 — elevated anti-nuclear antibody, asymptomatic
seroma (Injury, poisoning and procedural complications) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
lymphocyte count decreased (Investigations) | 1 | 0
anorexia (Metabolism and nutrition disorders) | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
dizziness (Nervous system disorders) | 1 | 2
headache (Nervous system disorders) | 5 | 3
tremor (Nervous system disorders) | 1 | 0
agitation (Psychiatric disorders) | 1 | 0
depression (Psychiatric disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
pain of skin (Skin and subcutaneous tissue disorders) | 1 | 2
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
other (Skin and subcutaneous tissue disorders) | 0 | 1
flushing (Vascular disorders) | 3 | 1
hot flashes (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No